CLINICAL TRIAL: NCT04056949
Title: The Efficacy and Safety of IBI308 Combined With Paclitaxel/Albumin-Bound Paclitaxel as Second-Line Therapy in Treating Patients With Extensive-Stage Small Cell Lung Cancer That Relapsed After Failing to Platinum-Etoposide Chemotherapy
Brief Title: Efficacy and Safety of IBI308 and Paclitaxel/Albumin Paclitaxel for SCLC Patients Who Failed Etoposide Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Junling Li (Other)
Responsible Party: Sponsor-Investigator, Junling Li, Clinical Professor, Peking Union Medical College
Organization: Peking Union Medical College (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC1977
Record Dates: First submitted 2019-08-09; First posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Extensive-Stage Small Cell Lung Cancer
Keywords: SCLC
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Albumin-Bound Paclitaxel; sintilimab

STUDY DESIGN:
Intervention Model Description: SCLC patients who have failed platinum-etoposide chemotherapy
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- IBI308 + Paclitaxel/Albumin-Bound Paclitaxel (Other): IBI308 Combined with Albumin-Bound Paclitaxe
  Interventions: Drug: Paclitaxel/Albumin-Bound Paclitaxel; Drug: IBI308

INTERVENTIONS:
Drug: Paclitaxel/Albumin-Bound Paclitaxel — Paclitaxel 175mg/m2 IV on day 1of 21 days cycle ;Number of Cycles: 4-6; or Albumin-bound paclitaxel 130mg/m2 IV on day 1 and 8 of 21 days cycle ;Number of Cycles: 4-6;
Drug: IBI308 — IBI308 200mg IV infusion, every 3 weeks,until disease progress or intolerable toxicity,used up to 1 year (or 16 cycles)

SUMMARY:
This phase II trial studies how well IBI308 combined with paclitaxel/albumin-bound paclitaxel work in treating participants with small cell lung cancer after failing to platinum-etoposide chemotherapy.

DETAILED DESCRIPTION:
Primary objective :

To estimate progression free survival (PFS) probability of patient who recurrent SCLC treated with IBI308 combined with paclitaxel/abumin-bound paclitaxel following progression on platinum-etoposide chemotherapy.

Secondary Objectives:

I.To evaluate the objective remission rate (ORR), disease control rate. (DCR),durative time of remission ( DoR）and overall survival (OS) of IBI308 combined with paclitaxel/abumin-bound paclitaxel following progression on platinum-etoposide chemotherapy.

II.To evaluate the safety of IBI308 combined with paclitaxel/abumin-bound paclitaxel following progression on platinum-etoposide chemotherapy.

Exploratory Objectives To evaluate the correlation of biomarkers with efficacy and toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent;
2. Over 18 years old and below 70 years old;
3. Histologically confirmed small-cell lung cancer;
4. Extensive disease(ED) according to the criteria of the Veteran's Administration Lung Cancer Group: (disease extended is defined as a disease beyond hemi thorax and supraclavicular lymph node areas.);
5. ED-SCLC treated with platinum-etoposide chemotherapy ,followed by disease progression or recurrence.
6. Availability of a biomarker detection tissue biopsy is required;
7. Eastern Cooperative Oncology Group (ECOG) performance status 0~1;
8. Life expectancy of greater than 12 weeks;
9. Participants may have evaluable or measurable disease, defined as at least one lesion（no previous radiotherapy）that can be accurately measured in at least one dimension with spiral CT scan, MRI within the past 28 days;
10. Women of child-bearing potential and men must agree to use adequate contraception prior to initiation of therapy and until to 6 month after this study;
11. White blood cell ≥ 3.5 × 109/L, absolute neutrophil count ≥1.5 × 109/L, platelet ≥100× 109/L and hemoglobin ≥9.0 g/dL;
12. Aspartate transferase,alanine aminotransferase ≤ 2.5 x ULN except in case of liver metastases (5 x ULN); Total bilirubin ≤1.5 x ULN except in case of Gilbert syndrome (3.0 mg/dL); Albumin≥3 g/dL;
13. Serum creatinine ≤1.5×ULN OR creatinine clearance≥40 mL/min;
14. Lipase < 1.5 x ULN except in case of having no clinical or imaging evidence of pancreatitis; Amylase ≤1.5 x ULN except in case of having no clinical or imaging evidence of pancreatitis; Alkaline phosphatase (ALP) ≤ 2.5 ULN except in case of bone metastasis;

Exclusion Criteria:

1. Mixed lung cancer or other types of lung cancer;
2. Prior immunotherapy, included but not limited to cytotoxic T lymphocyte-associated antigen-4 (CTLA-4) inhibitors, PD-1 inhibitors, PD-L1/2 inhibitors or other drugs targeting T cells;
3. Received high-dose radiation therapy in thoracic field within the past 6 months, Dt (> 30 Gy);
4. Active or untreated central nervous system (CNS) metastases;
5. Patients with cytologically positive pleural, peritoneal or pericardial fluid are not eligible;
6. History of autoimmune disease.Patients with a history of hypothyroidism origin autoimmune treated with a stable dose replacement therapy may be eligible for this study. Patients with controlled type 1 diabetes treated with insulin are eligible in this study;
7. Corticosteroid with a daily dose over 10 mg prednisolone or other immunosuppressive agents were used within 14 days before the first cycle;
8. Patients should not receive a vaccine during the four weeks preceding the day 1 of cycle 1, and shall not receive a vaccine during the study;
9. Idiopathic pulmonary fibrosis history, radioactive pneumonia requiring steroid therapy, organizing pneumonia (eg, bronchiolitis obliterans), drug-induced lung disease, idiopathic pulmonary or active signs of pneumonia or interstitial lung infiltrate (any cause) detected on the lung scan selection;
10. History of active Bacillus Tuberculosis;
11. Except hair loss and fatigue, toxicities caused by previous anti-cancer therapies need to be restored to < CTCAE 4.03 grade 1 before starting treatment on protocol;
12. History of any one or more of the following conditions within the past 6 months:symptomatic peripheral vascular disease, pulmonary embolism or untreated deep venous thrombosis (DVT), cerebrovascular accident or transient ischemic attack;
13. History of any one or more of the following conditions within the past 6 months: gastrointestinal ulcer, gastrointestinal perforation, corrosive esophagitis or gastritis, inflammatory bowel disease or diverticulitis, abdominal fistula, tracheoesophageal fistula or abdominal abscess;
14. History of any one or more of the following cardiovascular conditions: Class III or IV congestive heart failure, as defined by the New York Heart Association; Unstable angina; Myocardial infarction within the past 6 months; Supraventricular or ventricular arrhythmia requires treatment or intervention;
15. Severe uncontrolled hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥ 100mmHg);
16. Tumors compress surrounding vital organs, such as the esophagus, with associated symptoms;
17. Uncontrolled hypercalcemia;
18. History of allergic reactions attributed to compounds of similar chemical or biologic composition to monoclonal antibody;
19. Prior malignancy. Note: Patients who have had another malignancy and were treated more than 5 years ago and have since been considered cured, or patients with a history of basocellular skin carcinoma or in situ carcinoma of the uterine cervix are eligible;
20. Mental illness, alcoholism, inability to quit smoking, drug abuse or drug abuse;
21. History of human immunodeficiency virus infection or has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C Virus (HCV) (e.g., HCV RNA is detected).
22. Pregnant or lactating female;
23. Any type of systemic anticancer therapy (chemotherapy or experimental drugs) within 4 weeks of starting treatment on protocol;
24. Other situations judged by researchers;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-08-05 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 12 months

SECONDARY OUTCOMES:
overall survival (OS) | 12 months
disease control rate (DCR) | 12 months
durative time of remission ( DoR） | 12 months
objective remission rate (ORR) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Junling Li, doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Junling Li, Beijing, Beijing Municipality, China